CLINICAL TRIAL: NCT06899828
Title: Unraveling Mechanism of Action of Extracorporeal Photopheresis in Heart and Lung Transplant Patients
Acronym: URRAH
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Claudia Del Fante, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: URRAH
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Heart Transplanted Patients; Lung Transplanted Patients; Chronic Lung Allograft Dysfunction (CLAD); Cardiac Allograft Vasculopathy
Keywords: ECP, heart and lung rejection, miRNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lung transplanted patients who receive diagnosis of chronic lung allograft dysfunction (CLAD)
- Heart transplanted patients who receive diagnosis of cardiac allograft vasculopathy (CAV)

SUMMARY:
This is a prospective observational single center national study. Lung and heart transplant patients with a definite diagnosis of chronic lung allograft dysfunction (CLAD) or cardiac allograft vasculopathy (CAV) will be assigned for extracorporeal photopheresis (ECP) as per common clinical practice to a 6-month ECP cycle with the aim of limiting progression of organ dysfunction. The exact mechanisms of ECP in chronic rejection after lung and heart transplantation (CLAD and CAV) are elusive but it is thought to induce apoptosis of lymphocytes and to generate regulatory T cells, which modulate transplant immune rejection by a complex effect.

DETAILED DESCRIPTION:
The primary objective of the present study is to identify the biomarkers associated to response to ECP after 6 months of treatment.

ELIGIBILITY:
Lung transplanted patients will be enrolled according to current per center protocol at diagnosis of established CLAD grade 1-2 (diagnosis will be made according to published guidelines) . Rate of graft function decline will be classified as rapid (>/= 100 ml/month) or slow (< 100ml/month) during the 6 months preceding ECP treatment. All patients will be diagnosed as CLAD after a failure of a 3-month trial with azithromycin. They will be enrolled in ECP treatment at CLAD grade 1-2. ECP response will be assessed after 6 months of treatment and patients experiencing > 10% decline with respect to baseline value at ECP initiation in graft function will be classified as non-responders.Heart transplanted patients with demonstrated CAV in a recent angiography (<6 months) in absence of acute cellular or antibodies mediated rejection at myocardial biopsy, will be enrolled The diagnosis of CAV will require the presence of thickening of the arterial intima in any epicardial artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart and lung transplant patients who receive diagnosis of chronic lung allograft dysfunction (CLAD) or cardiac allograft vasculopathy (CAV)
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
identification the primary mechanism of action of ECP in CLAD and CAV by analyzing biological markers (such as relative expression levels of microRNAs, potentially involved in immune regulation), associated to response to a 6 month-ECP treatment course | After 6 months from ECP treatment

SECONDARY OUTCOMES:
Correlation between up-regulation or down-regulation of miRNAs at 6 months of therapy respect to baseline and other immune variables (regulatory T cells activation and differentiation, inflammatory cytokines levels and presence of anti-HLA antibodies) | After 6 months of therapy
Evaluation the effectiveness of ECP | After 2 years of follow-up from ECP
  Evaluation the effectiveness of ECP in reducing cardiovascular mortality and preventing percutaneous myocardial revascularization and hospitalization by cardiovascular causes at 2 years of follow-up in comparison to a control population of heart transplant recipients with CAV included in our historical archive
Effect of ECP on progression of myocardial fibrosis evaluated at CMR | After 6 months of treatment
Effect of ECP on ventricular function evaluated at echocardiography | After 6 months of treatment
Trend of heart failure biomarkers (NT proBNP or BNP) after 6 months of treatment | After 6 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy